CLINICAL TRIAL: NCT00166959
Title: Reliability and Validity of Modified Postural Assessment Scale for Stroke Patients and the Application of This Scale on Early Detection of Patients With Stroke at High Risk of Falls
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700931
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-06

CONDITIONS: Stroke
Keywords: Stroke patients; Falls; Reliability; Validity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purposes of this study are to investigate the reliability and validity of the modified Postural Assessment Scale for Stroke Patients (mPASS) and its applications in early detection of fall-prone patients.

The intraclass correlation coefficient will be used to examine the intra-rater reliability, inter-rater reliability, and the Cronbach's alpha will be used to examine the internal consistency of the 16 items of mPASS.

DETAILED DESCRIPTION:
Due to the impaired balance function, patients with stroke show high incidence of falls. Impaired postural stability has been shown as one of the primary risk factors of falls in these patients. Research has shown that patients who have moderate level of mobility and stability are more likely to fall than those who have very good or very poor mobility and stability. Therefore, there is an urgent need for physical therapists, who are used to play an important role in improving balance function of patients with stroke, to be able to early detect stroke patients who are at high risk of falls, and to implement fall prevention training and education on these patients. However, to date, there is not any clinical assessment scale that can be used for early detection of fall-prone stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* between 30 and 80 years old
* first onset or recurrent stroke as a result of a single cerebral vascular accident (ischemic or hemorrhage stroke)
* ever received medical or rehabilitation therapies at National Taiwan University Hospital
* being willing to take the clinical assessments and accept the vedio record

Exclusion Criteria:

* having unstable vital sign, unconsciousness, or having serious cognitive, perception, and language impairment, and being unable to follow the order of the experimenter
* having other neurological diseases(ex. Parkinson's disease or cerebellar disease etc.), or moderate to severe neuromuscular or musculoskeletal disorders, or disorders from systematic diseases those will influence the balance performance other than stroke

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2005-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Chein-Wei Chang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan